CLINICAL TRIAL: NCT00484510
Title: A Randomized, Placebo-controlled, Double Masked 120 Subject "Futility Design" Clinical Trial of Ascorbic Acid Treatment of Charcot Marie Tooth Disease Type 1A.
Brief Title: High Dose Ascorbic Acid Treatment of CMT1A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Muscular Dystrophy Association (Other); Charcot-Marie-Tooth Association (Other)
Responsible Party: Principal Investigator, Michael E. Shy, MD, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC074406MP2F; MDA4193
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Charcot-Marie-Tooth Disease, Type Ia
Keywords: Ascorbic Acid; Vitamin C; Charcot Marie Tooth; CMT; CMT1a
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ascorbic Acid (Experimental)
  Interventions: Drug: Ascorbic acid (Vitamin C)
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ascorbic acid (Vitamin C) — Eight 500 mg capsules/day of ascorbic acid. Subjects will take four (4)capsules each morning and four (4) capsules each evening for 24 months. (Total 4 gr/day).
  Arms: Ascorbic Acid
Drug: placebo — Eight 500 mg capsules/day of placebo. Subjects will take four (4)capsules each morning and four (4) capsules each evening for 24 months.
  Arms: Placebo

SUMMARY:
This study will look at the impact of ascorbic acid (Vitamin C) on the progression of disease in people with CMT1A as compared to volunteers receiving a placebo. This study will assess whether is it futile to proceed with a larger, longer-term, placebo-controlled study.

DETAILED DESCRIPTION:
Charcot Marie Tooth disease (CMT), or inherited peripheral neuropathies, are among the most frequent heritable disorders, affecting approximately 1 in 2500 people. The most frequent genetic form of CMT is CMT1A. CMT1A is caused by a 1.4 Mb duplication within chromosome 17p11.2 in the region containing the PMP22 gene. Most subjects with CMT1A have a "typical" phenotype characterized by onset in childhood or early adulthood, distal weakness, sensory loss, foot deformities and absent reflexes. How increased expression of PMP22 causes these disabilities is unknown but is currently being investigated in both animal and tissue culture systems. In this study, researchers will evaluate whether ascorbic acid (Vitamin C), administered orally, slows clinical progression of CMT1A and affects the PMP22 mRNA levels of myelinated peripheral nerve fibers obtained from biopsies of glabrous skin.

ELIGIBILITY:
Inclusion Criteria:

* The subject has CMT1A, defined by the duplication on chromosome 17p11.2 performed by either Pulse Field Gel Electrophoresis or Fluorescence In Situ Hybridization (FISH) by a CLIA certified laboratory, OR the subject has a first or second degree relative with a documented duplication performed by the above methods AND the subject has uniform motor conduction slowing of the median or ulnar nerve between 16 and 30 m/s.
* The subject is between 13 and 70 years of age.
* The subject, if 18 years or older, has signed the Informed Consent Form and agrees to follow the stipulations of the protocol.
* If the subject is less than 18, his or her parents or guardians have signed the Informed Consent Form and agree to follow the stipulations of the protocol. The subject has also signed a written assent form.

Exclusion Criteria:

* A known neuropathy from another source (For example, diabetes, drug induced, alcohol, etc.)
* The subject has ever received Vincristine.
* The subject has a known allergy to ascorbic acid.
* The subject has ever had kidney stones.
* The subject has a known history of G6PD deficit.
* The subject has a history of hemochromatosis.
* The subject suffers from a serious illness or medical condition that is not stabilized or that could require hospitalization.
* The subject has a high ascorbic acid level at screening.
* The subject is pregnant or nursing.
* The subject, in the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason.
* The subject participates to another clinical trial or is still within a washout period of a previous clinical trial.
* The subject is taking neurotoxic medications.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean change in the CMT Neuropathy Scale following high dose ascorbic acid ingestion, assessed at baseline and every 6 months throughout the trial. | 25 months per subject from baseline to completion.

SECONDARY OUTCOMES:
Evaluation of PMP22 mRNA levels of myelinated peripheral nerve fibers. | Baseline and Month 24.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Lewis, MD, Principal Investigator — Wayne State University, Dept. of Neurology
Locations (3):
- United States (3):
  - Johns Hopkins University, Dept of Neurology, Baltimore, Maryland
  - Wayne State University, Dept of Neurology, Detroit, Michigan
  - University of Rochester Medical Center, Dept of Neurology, Rochester, New York

REFERENCES:
- [Derived] Lewis RA, McDermott MP, Herrmann DN, Hoke A, Clawson LL, Siskind C, Feely SM, Miller LJ, Barohn RJ, Smith P, Luebbe E, Wu X, Shy ME; Muscle Study Group. High-dosage ascorbic acid treatment in Charcot-Marie-Tooth disease type 1A: results of a randomized, double-masked, controlled trial. JAMA Neurol. 2013 Aug;70(8):981-7. doi: 10.1001/jamaneurol.2013.3178. PMID 23797954